CLINICAL TRIAL: NCT03677167
Title: The Effect of Barefoot Walking on Pain Level, Functional Status and Pressure Pain Threshold in Patients With Plantar Chronic Heel Pain
Brief Title: The Effect of Barefoot Walking Plantar Chronic Heel Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meuhedet. Healthcare Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MeuhedetHCO
Record Dates: First submitted 2018-08-29; First posted 2018-09-19 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2019-12

CONDITIONS: Plantar Fascitis
Keywords: chronic plantar heel pain; barefoot; treadmill; Plantar Fascitis
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: The study will include 52 subjects with heel pain for more than 12 weeks. The subjects will be randomly assigned to one of two groups: a barefoot walking group on a treadmill and a walking group in shoes on a treadmill. The subjects will receive treatment twice a week at the Meuhedet Health Fund Institute for 4 weeks. All subjects will be instructed to walk on the treadmill until they reach level 6 on the Short Borg Scale. In addition, all subjects will receive an ultrasound treatment for 5 minutes each session. Before and after the intervention, the subjects will complete the SF-36 questionnaire, and will assess the level of pain they experience on the heel during initial treading down from the bed in the morning. In addition, the minimum pain threshold and pain tolerance will be checked with an algometer at relevant points in the heel and the speed and walking time will be documented.
Who Masked: Outcomes Assessor
Masking Description: The physiotherapist who examines patients before and after the intervention does not know which group the patient belongs to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- walking on a treadmill barefoot group (Experimental): 26 Patients in this group will walk barefoot on the treadmill and will be asked to walk barefoot at home and report the time of barefoot walking at home
  Interventions: Other: walking on a treadmill
- Walking on a treadmill with shoes group (Active Comparator): 26 Patients in this group will walk with shoes on the treadmill
  Interventions: Other: walking on a treadmill

INTERVENTIONS:
Other: walking on a treadmill — Patients will go on the treadmill (barefoot or with shoes) twice a week for a month, up to a medium-high level effort, and will receive ultrasound treatment for the painful heel spot
  Other Names: Ultrasound wave therapy

SUMMARY:
Many patients suffer from chronic heel pain, and studies have not yet found the most appropriate treatment. There are some researchers who claim that the pain is caused by weakness in the muscles of the foot, which causes increased pressure in the heel. In walking, the muscles of the foot are activated and strengthened. No research has yet been done on whether walking (barefoot or with shoes) on a treadmill reduces pain in the heel and improves function.

DETAILED DESCRIPTION:
A bare foot functions differently than a foot in a shoe while walking, as there are differences in movement, muscle tone, pressure and sensation. Wearing shoes over the years can cause changes in walking and pain. In the examination of the feet of patients suffering from chronic pain in the heel was found a smaller volume of muscle, and calcification in the heel area that could be caused by increased pressure. Although the trend of physiotherapy treatments has changed in recent years from passive to active treatments, the overwhelming majority of studies are testing passive therapies only as a treatment option for chronic heel pain. Barefoot walking has not been tested as an option for treating chronic pain in the heel, although there are studies indicating that bare feet lead to reduced heel pressure, increased muscle work, and better proprioception.The purpose of this study is to examine the effect of barefoot walking on the level of pain, function and pain threshold for stress in patients with chronic heel pain.

ELIGIBILITY:
Inclusion Criteria:

* Local pain in the heel that lasts more than 12 weeks,
* pain in the first steps in the morning
* Pain that disappears in situations of weightlessness
* Ability to walk on a moving track.

Exclusion Criteria:

* Pain in proximal areas along the leg or lower back pain that can radiate to the heel
* Sensory disorders for various reasons
* Tumors, fractures, previous operations in the lower extremities
* Irritable cardiovascular problems
* Balance problems and dizziness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
change in results of sf-36 scale from baseline to 4 weeks of intervention and 8 weeks | before intervention, after 4 weeks of intervention, after 4 weeks from the end of intervention (i.e. baseline to 4 weeks of intervention and 8 weeks)
  This is a questionnaire consisting of eight separate parts, each section examining a different aspect of quality of life. In the evaluation of pain in the heel, it is customary to use a part that assesses functional function, and in part that evaluates physical pain. The score ranges from 0 - very low, to 100 - very high. A change of 7.8 points indicates a change in the level of pain and physical function.

SECONDARY OUTCOMES:
change in results of VAS pain in the heel that appears on the first step in the morning from baseline to 4 weeks and 8 weeks | before intervention, after 4 weeks of intervention, after 4 weeks from the end of intervention (i.e. baseline to 4 weeks of intervention and 8 weeks)
  The ladder is 10 cm long, and the patient must surround the number that corresponds to his or her pain intensity, 0 - does not hurt at all, and 10 - the most severe and intolerable pain. When a change of 1.4 cm out of 10 cm indicates a change in the patient's pain level
change in results of Pain threshold severity for minimum pressure and tolerance threshold for pain for pressure at five points in the heel, from baseline to 4 weeks and 8 weeks | before intervention, after 4 weeks of intervention, after 4 weeks from the end of intervention (i.e. baseline to 4 weeks of intervention and 8 weeks)
  The algometer will measure the intensity of the pressure at the point of pain until reaching the minimum pain (P1) and also until reaching the threshold of pain tolerance
change in results of Three clinical tests to diagnose chronic pain in the heel, from baseline to 4 weeks and 8 weeks | before intervention, after 4 weeks of intervention, after 4 weeks from the end of intervention (i.e. baseline to 4 weeks of intervention and 8 weeks)
  Three clinical trials have been found to be relevant to the diagnosis of chronic heel pain. All the tests listed below are performed on the painful leg and until the first sensation of pain (p1) is produced:
  1. Static standing on one leg: measuring the number of seconds (up to 20 sec) and the level of pain on a visual analog scale (VAS);
  2. Crouching on one leg: measuring the number of repetitions (up to10 rep) and the level of pain according to VAS;
  3. Ascension on fingertips: Measuring the number of repetitions (up to10 rep) and the level of pain according to VAS.
  It was found that when pain is produced in one of the above tests, the patient may be diagnosed with chronic heel pain. The results options for all of the above tests are "positive" (if at least one of the tests creates pain) or "negative" (if non of the tests creates pain)
change in the duration (minuets) of walking on the treadmill until reaching level 6 on the short borg scale,from base line to 4 weeks | 1st intervention, after 4 weeks of intervention
  the duration of walking on the treadmill until reaching level 6 on the short borg scale.
change in the walking speed (Kilometer/hour) on the treadmill until reaching level 6 on the short borg scale,from baseline to 4 weeks | 1st intervention, after 4 weeks of intervention
  change in the walking speed (Kilometer/hour) on the treadmill until reaching level 6 on the short borg scale
short borg scale | 1st intervention, after 4 weeks of intervention
  The short borg scale is a scale that assesses the intensity of physical activity according to the subjective feeling of the patient. The short borg scale ranges from 0 - rest mode to 10 - maximum exertion.
  Training at level 5-6 has been found to be effective in achieving physiological improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Rael Strous, MD,MHA, Principal Investigator — Meuhedet Health Care
Locations (1):
- Meuhedet Health Care Phisiotherapy Clinic, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
Publication of the research in the university's databases and scientific journals
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2021
Access Criteria: After the thesis is completed, the research details will be available in the databases of Tel Aviv University, and after it is written as an article, it will be available in a journal that will publish the research